CLINICAL TRIAL: NCT05297110
Title: Efficacy of a Treatment Based on Olive Leaf Extracts in the Control of Cardiovascular Risk Factors
Brief Title: Olive Leaf Extracts in the Control of Cardiovascular Risk
Acronym: Atherolive
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, Head of Emergency departement, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Atherolive
Record Dates: First submitted 2021-11-17; First posted 2022-03-28 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Diabetes Mellitus, Type 2; Hypertension
Keywords: diabetes; hypertension; atherolive
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atherolive group (Active Comparator): In each study population, the patient will be assigned to one of two treatments (atherolive or placebo) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.
  Interventions: Drug: atherolive
- placebo group (Placebo Comparator): In each study population, the patient will be assigned to one of two treatments (atherolive or placebo) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.
  Interventions: Drug: atherolive

INTERVENTIONS:
Drug: atherolive — In each study population, the patient will be assigned to one of two treatments (atherolive or placebo) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.

SUMMARY:
This study will be carried out in 2 emergency departments (at the exit of the emergency room) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

Patients over 18 years of age with:

1. Arterial hypertension (hypertension).
2. Or diabetes.
3. Or one or more other cardiovascular risk factors (AHA, ESC) or risk of cardiovascular disease> 20% according to the Framingham scale (apart from hypertension and diabetes were included.

DETAILED DESCRIPTION:
This study will be carried out in 2 emergency departments (at the exit of the emergency room, patients included in the GR2 study) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

All the population will benifit of a biological assessment which include:

* Complete lipid profile, blood sugar, creatinine
* HbA1c (if the patient is diabetic).
* Inflammatory assessment: reactive protein C

Three populations will be randomized:

1. The population of patients with hypertension.
2. The population with diabetes.
3. The population of patients with other risk factors with a Framingham> 20% In each study population, the patient will be assigned to one of two treatments (atherolive or placebo). The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.

For patients in the hypertension group:

A blood pressure or glycemic holter will be carried out for 24 hours respectively and diabetics.

The raw data (hourly averages) are stored on a computer .

For diabetic patients:

Continuous blood glucose monitoring to measure indices of glycemic variability is performed at baseline. These patients will be equipped with an iPro continuous glycemic monitoring

For other patients (Framingham> 20%) For this group, the initial assessment will also include a specific assessment. Assessment of endothelial function by the digital plethysmography method to measure flow-mediated dilation (FMD or flow-mediated dilation expressed by the RHI) and specific biological assesement ( Willebrand factor, Homocystein )

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with:

  1. Arterial hypertension (hypertension).
  2. Or diabetes.
  3. Or one or more other cardiovascular risk factors (AHA, ESC) or risk of cardiovascular disease> 20% according to the Framingham scale (apart from hypertension and diabetes.

Criteria exclusion:

-. Exclusion criteria: None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
rate of blood pressure reduction | 90 days
  blood pressure reduction on 24 hours holter
rate of fasting glycemia level reduction | 90 days
  morning glycemic cycle

SECONDARY OUTCOMES:
rate of lipid balance variation The secondary endpoint (for the 3 study populations): lipid profile | 90 days
  variation in lipid balance
rate of hospitalization for cardiovascular disease | 90 days
  rate of hospitalization for cardiovascular disease: acute infarction, hypertension, acute stroke
rate of adverse effects | 90 days
  number of adeverse evnets reported

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Professor, Principal Investigator — University of Monastir
Locations (1):
- Fattouma Bourguiba Monastir University Hospital Center, Monastir, Tunisia